CLINICAL TRIAL: NCT03477474
Title: Registry of Guardant360® Use and Outcomes In People With Advanced Cancer
Acronym: GEODE
Status: Terminated | Type: Observational
Why Stopped: Alternative data published
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-MX-003
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Guardant Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to collect data that describes the characteristics of people with advanced cancer for whom the Guardant360 assay is ordered and to observe their clinical outcomes after receiving their results.

DETAILED DESCRIPTION:
This is a prospective, descriptive registry of people with advanced cancer for whom a Guardant360 assay has been ordered by their health care providers. The registry is divided into modules according to primary cancer diagnosis. Module 1 includes subjects with advanced NSCLC with additional modules added later in the study.

All eligible people for whom blood for a Guardant360 assay has been collected will be invited to participate in the registry. Subject demographics and relevant medical history will be collected at the time of enrollment. Information on tumor molecular testing, treatment decisions, and clinical outcomes from the time of enrollment will be collected in a prospective manner. The registry does not require any specific treatments or procedures but rather collects information on the treatment journey of each participant. Subjects may participate in other clinical studies while also participating in GEODE.

ELIGIBILITY:
General Inclusion Criteria:

1. 18 Years of age or older
2. Ability to provide written informed consent
3. Blood collected for the most recent Guardant360 test within 8 weeks prior to enrollment

General Exclusion Criteria

1. Pregnancy at the time of the qualifying Guardant360 blood collection
2. History of the allogeneic organ or tissue transplant

Module 1 (Non-Small Cell Lung Cancer)

Inclusion Criteria

1. NSCLC, confirmed by histology or cytology
2. Advanced disease, defined as: stage IIIB or IV NSCLC at the time of the qualifying Guardant360 blood collection; or for subjects with an initial diagnosis of Stage I-IIIA disease, NSCLC that is recurrent or metastatic at the time of the qualifying Guardant360 blood collection
3. One of the following conditions at the time of the qualifying Guardant360 blood collection:

   * No prior systemic therapy for advanced disease OR
   * All three of the following conditions:

1. A history of prior systemic therapy for advanced disease, 2. Disease progression within the previous four weeks, & 3. No new systemic therapy for advanced disease

Exclusion Criteria Subjects with a diagnosis or history of any cancer involving the lung that is not classified as NSCLC, including but not limited to small cell carcinoma, neuroendocrine or carcinoid tumor, lymphoma, mesothelioma, metastatic non-lung carcinoma, or cancer of unknown primary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Population Description:
  People With Advanced Cancer for whom the Guardant360 assay is ordered.
  Module 1 [NSCLC] Description:
  People with Advanced NSCLC for whom the Guardant360 assay is ordered.
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Estimate Progression Free Survival (PFS) | 24 Months

SECONDARY OUTCOMES:
Duration of treatment response | 24 Months
Time of tumor progression | 24 Months
time to treatment failure | 24 Months
Overall survival | 24 Months
Turnaround time for Guardant360 and tissue based genomic testing | 24 Months
Molecular alteration discovery rates for various alterations | 24 Months
Tumor response rates | 24 Months
Quantity not sufficient rescue rates | 24 Months
Tissue incomplete rescue rate | 24 Months
The rate at which treatment plans are changed following results of the Guardant360 test | 24 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Cross, Fort Lauderdale, Florida, United States